CLINICAL TRIAL: NCT00003063
Title: Adjuvant Chemoimmunotherapy for Colorectal Cancer
Brief Title: Biological Therapy With Combination Chemotherapy in Patients With Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Institute of Oncology (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065728; CNR-TONE-01; EU-97011
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2005-11

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage III colon cancer; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Interferon-alpha; Fluorouracil; Leucovorin; Levamisole

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: fluorouracil
Drug: leucovorin calcium
Drug: levamisole hydrochloride

SUMMARY:
RATIONALE: Biological therapies use different ways to stimulate the immune system and stop cancer cells from growing. Combining chemotherapy with biological therapy may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of treatment using levamisole with treatment using interferon alfa and combination chemotherapy consisting of fluorouracil and leucovorin in patients with stage II or stage III colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the efficacy of the addition of levamisole or alfa interferon to fluorouracil and leucovorin calcium (folinic acid) as an adjuvant treatment of intraperitoneal colorectal cancer.

OUTLINE: This is a three arm study. Patients are randomized to receive either levamisole, alfa interferon, or no treatment.

* Arm I: Patients receive levamisole PO for 3 days every 2 weeks for 6 months before and after surgery. Fluorouracil IV bolus and leucovorin calcium (folinic acid) IV over 1 hour are administered on days 1-5 every 4 weeks for 6 cycles after surgery.
* Arm II: Patients receive alfa interferon-2a SC on 3 alternate days for a week before surgery and for 6 months after surgery. Fluorouracil IV bolus and folinic acid IV over 1 hour are administered on days 1-5 every 4 weeks for 6 cycles after surgery.
* Arm III: Patients undergo surgery followed by fluorouracil IV bolus and folinic acid IV over 1 hour on days 1-5 every 4 weeks for 6 cycles.

Patients are followed every 3 months for 2 years, then every 6 months.

PROJECTED ACCRUAL: 350 patients per arm will be accrued for a total of 1,050 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage T3-T4 N0 or T1-T4 N1-3 colorectal cancer
* No evidence of residual disease after surgery
* Tumor located above peritoneal reflection
* No distant metastases

PATIENT CHARACTERISTICS:

Age:

* 75 and under

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* SGPT less than 2 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No serious cardiac ischemia

Other:

* Adequate metabolic functions
* No prior neoplasm
* No prior/concurrent illness
* No insulin-dependent diabetes

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy for the current cancer

Chemotherapy

* No prior chemotherapy for the current cancer

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for the current cancer

Surgery

* Not specified

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 1991-11

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Tonelli, MD, Study Chair — Universita Degli Studi di Florence - Policlinico di Careggi
Locations (85):
- George Papanicolaou General Hospital, Thessaloniki, Greece
- Italy (83):
  - Ospedale Bassini, Balsamo Cinisello
  - Universita Degli Studi di Bari Policlinico, Bari
  - Spedali Civili, Brescia
  - Cattedra di Oncologia Medica - Universita, Cagliari
  - Ospedale Oncologico A. Businco, Cagliari
  - Ospedale San Michele, Cagliari
  - Ospedale Sant Anna, Como
  - Ospedale Valduce, Como
  - Ospedale Di Conselice, Conselice
  - Ospedale Civile Cosenza, Cosenza
  - Ospedale Maggiore Crema, Crema
  - Ospedale Santa Croce, Cuneo
  - Ospedale Civile Feltre, Feltre
  - Universita di Ferrara, Ferrara
  - Universita Degli Studi di Firenze - Policlin. di Careggi, Firenze (Florence)
  - Policlinico di Careggi, Firenze (Florence)
  - U.S.L. 10 Villa Ognissanti, Florence
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa (Genova)
  - Ospedale San Martino/Cliniche Universitarie Convenzionate, Genoa (Genova)
  - Ospedale Galliera Oncologia, Genova (Genoa)
  - Ospedale Di Gorgonzola, Gorgonzola
  - Ospedale Legnago USSL 21, Legnago
  - Ospedale Maggiore Lodi, Lodi
  - Ospedale Umberto I, Lugo DI Romagna
  - U.S.S.L. 72 Magenta, Magenta
  - Carlo Poma Hospital, Mantova
  - Ospedale Di Predabissi Melegnano, Melegnano
  - Azienda USSL NO 8, Merate
  - Instituto Di Oncologia, Messina
  - Ospedale Civile Umberto I, Mestre
  - Ospedale San Giuseppe, Milan
  - Consorzio Provinciale Antitubercolare, Milan
  - Istituto Scientifico H.S. Raffaele, Milan
  - Istituto Di Science Biomediche San Paolo, Milan
  - Casa Di Cura San Ambrogio, Milan
  - Ospedale San Carlo Borromeo, Milano (Milan)
  - Ospedale Luigi Sacco, Milano (Milan)
  - Ospedale Maggiore Ca Granda, Milano (Milan)
  - Ospedale Santa Croce, Moncalieri
  - Nuovo Ospedale San Gerardo, Monza
  - Ospedale Civile Asilo Vittoria, Mortara
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples
  - Federico II University Medical School, Naples (Napoli)
  - Istituto Tumori/Fondazione Pascale, Naples (Napoli)
  - Ospedale Vincenzo Monaldi, Napoli
  - Ospedale C. Ascalesi, Napoli
  - Ospedale Civile Negrar, Negrar
  - Azienda Ospedaliera di Padova, Padova (Padua)
  - University of Padua, Padua
  - Ospedale Civico E Benefratelli, Palermo
  - Ospedale Maggiore Parma, Parma
  - Ospedale Torrette University Ancona, Parma
  - Ospedale Silvestrini, Perugia
  - Ospedale Agnelli, Pinerolo
  - Ospedale Sta. Maria Delle Croci, Ravenna
  - Azienda Ospedaliera, Reggio Emilia
  - Ospedale Civile Rho, Rho
  - Istituti Fisioterapici Ospitalieri - Roma, Rome
  - Ospedale San Filippo Neri, Rome
  - Ospedale Carlo Forlanini, Rome
  - Ospedale S. Camillo-Forlanini, Rome
  - Azienda Policlinico Umberto Primo, Rome
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
  - Policlinico Militare Celio, Rome
  - ASL NO. 1 Imperiese, Sanremo
  - Azienda USSL No 4, Saronno
  - Istituto Clinica Medica, Sassari
  - Ospedale S.S. Annunziata, Savigliano
  - Ospedale Sesto San Giovanni, Sesto San Giovanni
  - Azienda Ospedaliera S. Maria, Terni
  - Ospedale Generale Prov. Boldrini, Thiene
  - Dispensario Igiene Sociale, Toino
  - Clinica Universita, Torino
  - Universita Torino, Torino
  - Ospedale S. Chiara, Trento
  - Ospedale San Isidoro, Trescore Balneario
  - Ospedale General Regional Ca Foncello, Treviso
  - Ospedale Maggiore dell' Universita, Trieste
  - Ospedale Cattinara, Trieste
  - Cattedra di Immunologia Clinica, Turin (TO)
  - Universita Degli Studi di Udine, Udine
  - Ospedale di Circolo e Fondazione Macchi, Varese
  - Ospedale San Bortolo, Vicenza
- Inha University Hospital, Incheon, South Korea